CLINICAL TRIAL: NCT06326892
Title: Postoperative Outcomes of Natural Orifice Specimen Extraction (NOSE) in Low Rectal Cancer Surgery
Brief Title: Natural Orifice Specimen Extraction in Low Rectal Cancer Surgery
Acronym: NOSES
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CHR1-101-2024
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Rectal Cancer; Surgery
Keywords: Rectal Cancer; Natural Orifice Specimen Extraction; Propensity score matched
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural Orifice Specimen Extraction (NOSE): Patients with low rectal cancer who underwent rectal resection with Natural Orifice Specimen Extraction (NOSE)
  Interventions: Procedure: Natural Orifice Specimen Extraction (NOSE)
- Controls: Patients with low rectal cancer who underwent rectal resection with traditional specimen extraction
  Interventions: Procedure: Traditional specimen extraction

INTERVENTIONS:
Procedure: Natural Orifice Specimen Extraction (NOSE) — Low rectal cancer resection with Total Mesorectal Excision (TME) and Natural Orifice Specimen Extraction (NOSE)
  Groups: Natural Orifice Specimen Extraction (NOSE)
Procedure: Traditional specimen extraction — Low rectal cancer resection with Total Mesorectal Excision (TME) and specimen extraction through Pfannenstiel incision
  Groups: Controls

SUMMARY:
This study aims to compare the postoperative outcomes of low rectal cancer patients who underwent surgery with Natural Orifice Specimen Extraction (NOSE) versus traditional Pfannenstiel extraction.

DETAILED DESCRIPTION:
Natural Orifice Specimen Extraction (NOSE) in colorectal surgery allows the extraction of the surgical specimen through the anal orifice. Several studies demonstrated improved postoperative pain, bowel movements, patient-reported cosmetic satisfaction, and psychological wellbeing after NOSE compared with traditional Pfannenstiel extraction. However, most of these studies focused on colon surgery. The aim of this retrospective propensity score matched study is to investigate the postoperative outcomes of NOSE in low rectal cancer surgery, classified according to the English National Low Rectal Cancer Development Programme (LOREC).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing low anterior resection with Total Mesorectal Excision (TME) for low rectal cancer between January 2017 and January 2023
* Patients with rectal cancer classified as "low" according to the English National Low Rectal Cancer Development Programme (LOREC)

Exclusion Criteria:

* Patients undergoing non-restorative procedures
* Patients undergoing immediate or delayed handsewn coloanal anastomosis
* Patients undergoing planned open surgery or unplanned conversion from minimally invasive to open surgery
* Patients with a concomitant diagnosis of Inflammatory Bowel Disease (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low rectal cancer to the English National Low Rectal Cancer Development Programme (LOREC) who underwent low rectal resection with Total Mesorectal Excision (TME)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infections (SSI) | 30 days after surgery
  Rate difference of 30-day Surgical Site Infections (SSI)- defined according to the definition of the Center for Disease Control and Prevention (CDC) [Ref]- between the study cohorts.

SECONDARY OUTCOMES:
Opioid rescue | From the date of surgery to the date of discharge
  Difference in the proportion of patients requiring opioid rescue during the hospitalization
Postoperative pain | 72 hours after surgery
  The median difference of 72-hour patient-reported pain- measured on the Visual Rating Scale (VRS)
Postoperative ileus | 30 days after surgery
  Rate difference of 30-day postoperative functional ileus (define as the absence of bowel function for at least three days)
Incisional hernia | 6 months after surgery
  The rate difference of six-month incisional hernia
Overall postoperative complications | 30 days after surgery
  The rate difference of overall 30-day postoperative complications, classified according to the Clavien-Dindo scale [ranging from 0 (no complications) to 5 (complications leading to death)]

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — IRCCS Huamanitas Research Hospital
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy